CLINICAL TRIAL: NCT00108004
Title: A Phase 3B, Multicenter, Open-Label Study Investigating the Clinical Utility and Safety of Pramlintide in Subjects With Type 1 and Type 2 Diabetes Mellitus Who Have Not Achieved Glycemic Targets With Insulin Therapy
Brief Title: Clinical Utility and Safety of Pramlintide in Subjects With Type 1 and Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 137-155
Record Dates: First submitted 2005-04-12; First posted 2005-04-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: Diabetes; Amylin; Symlin; pramlintide acetate
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — pramlintide

ARMS (1):
- Pramlintide (Experimental): Pramlintide acetate injection is a clear, colorless, sterile solution for SC injection.
  It consists of pramlintide in sodium acetate buffer, pH 4.0, containing 43-mg/mL mannitol as an iso-osmolality modifier and 2.25 mg/mL metacresol as a preservative
  Interventions: Drug: pramlintide acetate

INTERVENTIONS:
Drug: pramlintide acetate — Pramlintide (0.6 mg/mL) in 5.0-mL multiple-draw glass vials for SC injection for 12weekes and after Pramlintide (1.0 mg/mL) 1.5 mL pen-cartridge. Subjects who do not switch to the pen-cartridge device at Week 12 will continue to administer pramlintide using a syringe and vial.

SUMMARY:
This open-label, multicenter study is designed to investigate the clinical utility and safety of pramlintide treatment in subjects with type 1 and type 2 diabetes who are failing to achieve the desired level of glycemic control using insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a clinical diagnosis of type 1 diabetes mellitus requiring treatment with insulin for a minimum of 6 months at Screening; -OR- The subject has a clinical diagnosis of type 2 diabetes requiring treatment with insulin with or without oral antidiabetic agents for a minimum of 6 months at Screening.
* The subject has a HbA1c of 7.0% to 11.0% at Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2003-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To investigate the clinical utility and safety of pramlintide in subjects with type 1 and type 2 diabetes mellitus | 6 months
  To investigate the clinical utility (change in HbA1c, seven-point glucose profile, body weight, and insulin use) and safety of pramlintide in subjects with type 1 and type 2 diabetes mellitus who have not achieved glycemic targets with insulin therapy.
Understand management issues in subjects with type 1 and type 2 diabetes mellitus | 6 months
  To collect data regarding the selection of subjects for pramlintide administration by healthcare professionals and to further understand management issues in subjects with type 1 and type 2 diabetes mellitus who have not achieved glycemic targets with insulin therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (48):
- United States (48):
  - Research Site, Anaheim, California
  - Research Site, Escondido, California
  - Research Site, La Jolla, California
  - Research Site, Los Gatos, California
  - Research Site, San Francisco, California
  - Research Site, Torrance, California
  - Research Site, New Britain, Connecticut
  - Research Site, Norwalk, Connecticut
  - Research Site, Norwich, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Clearwater, Florida
  - Research Site, Orlando, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Idaho Falls, Idaho
  - Research Site, Indianapolis, Indiana
  - Research Site, Vincennes, Indiana
  - Research Site, Topeka, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Bloomfield Hills, Michigan
  - Research Site, Tupelo, Mississippi
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Moorestown, New Jersey
  - Research Site, Neptune City, New Jersey
  - Research Site, Roseland, New Jersey
  - Research Site, New York, New York
  - Research Site, Williston Park, New York
  - Research Site, Yonkers, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Lakewood, Ohio
  - Research Site, Westlake, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Wilkes-Barre, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Sumter, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Dallas, Texas
  - Research Site, Olympia, Washington
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Herrmann K, Frias JP, Edelman SV, Lutz K, Shan K, Chen S, Maggs D, Kolterman OG. Pramlintide improved measures of glycemic control and body weight in patients with type 1 diabetes mellitus undergoing continuous subcutaneous insulin infusion therapy. Postgrad Med. 2013 May;125(3):136-44. doi: 10.3810/pgm.2013.05.2635. PMID 23748514
- [Derived] Karl D, Philis-Tsimikas A, Darsow T, Lorenzi G, Kellmeyer T, Lutz K, Wang Y, Frias JP. Pramlintide as an adjunct to insulin in patients with type 2 diabetes in a clinical practice setting reduced A1C, postprandial glucose excursions, and weight. Diabetes Technol Ther. 2007 Apr;9(2):191-9. doi: 10.1089/dia.2006.0013. PMID 17425446
- [Derived] Edelman SV, Darsow T, Frias JP. Pramlintide in the treatment of diabetes. Int J Clin Pract. 2006 Dec;60(12):1647-53. doi: 10.1111/j.1742-1241.2006.01187.x. PMID 17109671